CLINICAL TRIAL: NCT04944433
Title: Safety and Efficacy of the Coronavirus Disease 2019 Vaccine in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Ministerio de Salud de Ciudad Autónoma de Buenos Aires (Other Government); University of Buenos Aires (Other)
Responsible Party: Principal Investigator, GUILLERMO JAVIER ROSA DIEZ, Principal investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 7412
Record Dates: First submitted 2021-06-18; First posted 2021-06-29 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Coronavirus Disease 2019 Vaccines; Renal Dialysis
Keywords: Seroepidemiologic Studies; Renal Dialysis; Coronavirus disease 2019 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is unknown whether Coronavirus disease 2019 vaccines confer the same high level of protection in patients with kidney disease as reported for participants in recent trials, who were generally healthy. Objectives: To evaluate the safety and efficacy of Coronavirus disease 2019 vaccines in hemodialysis patients.

DETAILED DESCRIPTION:
Given the vulnerability of people with chronic kidney disease to Coronavirus 2019 , leading nephrology societies such as the National Kidney Federation and the American Kidney Foundation have issued statements calling for prioritization of these patients for vaccination. It is unknown whether Coronavirus disease 2019 vaccines confer the same high level of protection in patients with kidney disease as reported for participants in recent trials, who were generally healthy.

Objectives:

1. Estimate the proportion of hemodialysis patients who present events supposedly attributed to vaccines and immunizations after having received a Coronavirus disease 2019 vaccine
2. Determine the levels of Immunoglobulin G antibodies in patients who received a Coronavirus disease 2019vaccine between the time before the first dose, at 21 days, at 40 days and at 120 days after immunization.

Methods Design: Multicenter, observational and analytical study of a prospective cohort of hemodialysis patients 18 years and older who received immunization with a Coronavirus disease 2019 vaccine in the Autonomous City of Buenos Aires in a vaccination plan.

Analysis The proportion of patients with Adverse events presumably attributable to vaccination and immunization will be estimated with its 95% confidence interval. The immunoglobulin G titer for coronavirus type 2 causing severe acute respiratory syndrome will be compared using Generalized Estimating Equations models.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age on hemodialysis in an immunization plan with a Coronavirus disease 2019 vaccine.

Exclusion Criteria:

* Contraindication to receive the vaccine.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients in an immunization plan with a COVID-19 vaccine from the hemodialysis centers of the Autonomous City of Buenos Aires
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Estimate the proportion of hemodialysis patients who present events supposedly attributed to vaccines and immunizations after having received a Coronavirus disease 2019 vaccine | one year
  Estimate the proportion of hemodialysis patients who present events supposedly attributed to vaccines and immunizations after having received a Coronavirus disease 2019 vaccine
To assess the change in the levels of Immunoglobulin G (IgG) antibodies from baseline at 21 days, at 40 days and at 120 days after immunization | one year
  To assess the change in the levels of Immunoglobulin G (IgG) antibodies from baseline at 21 days, at 40 days and at 120 days after immunization

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo IP Rosa Diez, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Jorge SI Geffner, Study Chair — University of Buenos Aires; Fernando SI Lombi, Study Chair — Sociedad Argentina de Nefrología; Marina SI Papaginovic, Study Chair — Sociedad Argentina de Nefrología; Ricardo SI Heguilen, Study Chair — Sociedad Argentina de Nefrología; Luciana Fernandez SI Paganti, Study Chair — Sociedad Argentina de Nefrología; Soledad SI Crucelegui, Study Chair — Hospital Italiano de Buenos Aires; Vanina SI Pagotto, Study Chair — Hospital Italiano de Buenos Aires
Locations (1):
- Universidad de Buenos Aires Facultad de Medicina, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Logunov DY, Dolzhikova IV, Zubkova OV, Tukhvatullin AI, Shcheblyakov DV, Dzharullaeva AS, Grousova DM, Erokhova AS, Kovyrshina AV, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Lubenets NL, Egorova DA, Shmarov MM, Nikitenko NA, Morozova LF, Smolyarchuk EA, Kryukov EV, Babira VF, Borisevich SV, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine in two formulations: two open, non-randomised phase 1/2 studies from Russia. Lancet. 2020 Sep 26;396(10255):887-897. doi: 10.1016/S0140-6736(20)31866-3. Epub 2020 Sep 4. PMID 32896291
- [Result] Logunov DY, Dolzhikova IV, Shcheblyakov DV, Tukhvatulin AI, Zubkova OV, Dzharullaeva AS, Kovyrshina AV, Lubenets NL, Grousova DM, Erokhova AS, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Egorova DA, Shmarov MM, Nikitenko NA, Gushchin VA, Smolyarchuk EA, Zyryanov SK, Borisevich SV, Naroditsky BS, Gintsburg AL; Gam-COVID-Vac Vaccine Trial Group. Safety and efficacy of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine: an interim analysis of a randomised controlled phase 3 trial in Russia. Lancet. 2021 Feb 20;397(10275):671-681. doi: 10.1016/S0140-6736(21)00234-8. Epub 2021 Feb 2. PMID 33545094
- [Result] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Result] Di Pasquale A, Bonanni P, Garcon N, Stanberry LR, El-Hodhod M, Tavares Da Silva F. Vaccine safety evaluation: Practical aspects in assessing benefits and risks. Vaccine. 2016 Dec 20;34(52):6672-6680. doi: 10.1016/j.vaccine.2016.10.039. Epub 2016 Nov 8. PMID 27836435
- [Result] Herve C, Laupeze B, Del Giudice G, Didierlaurent AM, Tavares Da Silva F. The how's and what's of vaccine reactogenicity. NPJ Vaccines. 2019 Sep 24;4:39. doi: 10.1038/s41541-019-0132-6. eCollection 2019. PMID 31583123
- [Result] Mitchell TC, Casella CR. No pain no gain? Adjuvant effects of alum and monophosphoryl lipid A in pertussis and HPV vaccines. Curr Opin Immunol. 2017 Aug;47:17-25. doi: 10.1016/j.coi.2017.06.009. Epub 2017 Jul 17. PMID 28728074
- [Result] Windpessl M, Bruchfeld A, Anders HJ, Kramer H, Waldman M, Renia L, Ng LFP, Xing Z, Kronbichler A. COVID-19 vaccines and kidney disease. Nat Rev Nephrol. 2021 May;17(5):291-293. doi: 10.1038/s41581-021-00406-6. Epub 2021 Feb 8. PMID 33558753
- [Result] Heldman MR, Limaye AP. SARS-CoV-2 Vaccines in Kidney Transplant Recipients: Will They Be Safe and Effective and How Will We Know? J Am Soc Nephrol. 2021 May 3;32(5):1021-1024. doi: 10.1681/ASN.2021010023. Epub 2021 Mar 24. No abstract available. PMID 33762353
- [Result] Scharpe J, Evenepoel P, Maes B, Bammens B, Claes K, Osterhaus AD, Vanrenterghem Y, Peetermans WE. Influenza vaccination is efficacious and safe in renal transplant recipients. Am J Transplant. 2008 Feb;8(2):332-7. doi: 10.1111/j.1600-6143.2007.02066.x. Epub 2007 Dec 19. PMID 18162092
- [Result] Labriola L, Scohy A, Seghers F, Perlot Q, De Greef J, Desmet C, Romain C, Morelle J, Yombi JC, Kabamba B, Rodriguez-Villalobos H, Jadoul M. A Longitudinal, 3-Month Serologic Assessment of SARS-CoV-2 Infections in a Belgian Hemodialysis Facility. Clin J Am Soc Nephrol. 2021 Apr 7;16(4):613-614. doi: 10.2215/CJN.12490720. Epub 2020 Nov 18. No abstract available. PMID 33208402
- See also: World Health Organization.Coronavirus disease 2019 vaccines. — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/covid-19-vaccines
- See also: Emergency registration of the product "Coronavirus disease 2019 Vaccine AstraZeneca". 2020. Argentina — https://www.argentina.gob.ar/noticias/registro-de-emergencia-del-producto-covid-19-vacuna-astrazeneca
- See also: Ministry of Health, Argentina. Strategic Plan for vaccination against Coronavirus disease 2019 in Argentina 2020 — https://www.argentina.gob.ar/sites/default/files/coronavirus-vacuna-plan-estrategico-vacunacion-covid-19-diciembre-2020.pdf
- See also: Ministry of Health, Argentina. Integrated Argentine Health Information System. 2020. — https://sisa.msal.gov.ar/sisadoc/docs/050203/nomivac_home.jsp